CLINICAL TRIAL: NCT05811897
Title: Un Meilleur Sommeil Pour Une Meilleure résilience : Une Plateforme en Ligne autogérée Pour Les Victimes d'Agression Sexuelle
Brief Title: RESILIENT : A Self-Managed Online Platform for Victims of Sexual Assault
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ministère de la Justice, Québec (Unknown)
Responsible Party: Principal Investigator, Geneviève Belleville, Full Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-409
Record Dates: First submitted 2023-02-10; First posted 2023-04-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder; Insomnia Disorder; Major Depressive Disorder
Keywords: mental health; post-traumatic stress disorder; psychological distress; sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Managed Online Treatment (Experimental): Participants manage their treatment online without the assistance of a therapist.
  Interventions: Behavioral: Self-Managed Online Treatment
- Therapist-Assisted Online Treatment (Active Comparator): Participant will be assisted through the process by a therapist who will provide support and encouragement for 15-20 minutes of contact per week for the duration of the treatment. Supportive contacts are not psychotherapy. They are intended to answer questions about the content of the platform, to review adherence to the exercises and to provide encouragement; they also allow for the rapid identification and referral of participants in case of need (e.g., suicidal crisis).
  Interventions: Behavioral: Therapist-Assisted Online Treatment

INTERVENTIONS:
Behavioral: Self-Managed Online Treatment — Self-help online cognitive-behavioural therapy focusing on post-traumatic stress, sleep and mood. The content is divided into three modules :
  * Coping with my trauma: psychoeducation about PTSD, cognitive restructuring prolonged exposure to avoided situations and memories (14 sessions)
  * Sleeping better: psychoeducation about, sleep management strategies (restriction of time in bed, stimulus control, sleep hygiene education), Imagery Rehearsal Therapy (10 sessions)
  * Improving my mood: psychoeducation about depression, behavioural activation; relaxation and mindfulness exercises; problem-solving strategies (6 sessions)
  A small portion of material is unlocked each week, and access to one module will be accessible after the completion of a previous one. Access to the online material will be unlimited in time. Participants complete self-report questionnaires after each module, the platform then provides feedback and suggests corresponding modules.
  Arms: Self-Managed Online Treatment
Behavioral: Therapist-Assisted Online Treatment — Same online intervention. Supervised graduate psychology students will provide brief regular weekly contacts for up to 30 weeks by video chat or phone, according to the participant's preference.
  Arms: Therapist-Assisted Online Treatment

SUMMARY:
There are 636,000 self-reported cases of sexual assault annually in Canada, and nine out of ten persons who have experienced sexual assault are women. Cognitive and behavioural therapies (CBT) are the treatment of choice for many psychological problems arising from sexual assault. However, accessing CBT is a significant challenge, especially for women who have experienced sexual assault who may be ashamed and not disclose the sexual assault. Online CBT is an effective option to circumvent these barriers. In addition to being accessible and less resource-intensive, studies report that patients are less inhibited and that the online environment provides greater emotional safety. There is also a growing body of evidence that online CBT programs requiring little or no contact with a mental health professional are effective, this having been demonstrated primarily with individuals with anxiety and mood disorders. But when it comes to treating the psychological symptoms of sexual assault in potentially vulnerable individuals, can we really suggest a self-care approach? There is no direct empirical evidence to support such a recommendation, and it is this important question that this project wishes to address. To compare the effectiveness, acceptability and user engagement in a self-managed treatment platform with or without the support of a therapist to reduce post-traumatic symptoms, depression and insomnia in people who have suffered one or more sexual assaults, 204 victims of sexual assault experiencing significant distress will be recruited and randomly assigned to either the self-managed or the therapist-assisted online treatment condition. Participants will complete measures assessing post-traumatic stress disorder, insomnia, depression, anxiety, and maladaptive beliefs before, during, after and 3 months after treatment. Secondary outcome will be and appreciation of the online treatment measures by a self-report questionnaire and a semi-structured interview. If effective in reducing symptoms, this treatment would offer the potential to support a self-care approach to treating a wide range of psychological symptoms resulting from sexual assault. The self-managed online platform would fill a service gap deplored by this population.

DETAILED DESCRIPTION:
Background. There are 636,000 self-reported cases of sexual assault annually in Canada, and nine out of ten persons who have experienced sexual assault are women. An alarming paradox is that although they suffer significant adverse consequences of sexual assault on their functioning, they have less social support than victims of other traumatic events to manage the psychological consequences of sexual assault. Cognitive and behavioural therapies (CBT) are the treatment of choice for many psychological problems arising from sexual assault. However, accessing CBT is a significant challenge, especially for women who have experienced sexual assault who may be ashamed and not disclose the sexual assault. Online CBT is an effective option to circumvent these barriers. In addition to being accessible and less resource-intensive, studies report that patients are less inhibited and that the online environment provides greater emotional safety. There is also a growing body of evidence that online CBT programs requiring little or no contact with a mental health professional are effective, this having been demonstrated primarily with individuals with anxiety and mood disorders. But when it comes to treating the psychological symptoms of sexual assault in potentially vulnerable individuals, can we really suggest a self-care approach? There is no direct empirical evidence to support such a recommendation, and it is this important question that this project wishes to address.

Objectives. To compare the effectiveness of the use of a self-managed treatment platform with or without the support of a therapist to reduce post-traumatic symptoms, depression and insomnia in people who have suffered one or more sexual assaults, to document the acceptability of the platform and user engagement in the platform.

Method. For this study, 204 victims of sexual assault experiencing significant distress will be recruited. Of these participants, 102 will be randomly assigned to the self-managed online treatment condition and 102 participants will be randomly assigned to the therapist-assisted online treatment condition. Both conditions will have access to the same online platform (RESILIENT) that contains modules addressing the reduction of post-traumatic stress, insomnia, and depression symptoms, as well as nightmares. The duration of the online treatment is flexible and can last up to 25 weeks.

Data analyses. Primary outcome are post-traumatic stress disorder, insomnia, depression and anxiety measured by self-report questionnaires assessing participants' symptoms completed before, during and 3 months after treatment. Secondary outcome will be maladaptive beliefs and appreciation of the online treatment measures by a self-report questionnaire and a semi-structured interview.

Foreseen impacts. If effective in reducing symptoms, this treatment would offer the potential to support a self-care approach to treating a wide range of psychological symptoms resulting from sexual assault. The self-managed online platform would fill a service gap deplored by this population.

ELIGIBILITY:
Inclusion Criteria:

1. Identify at least in part as a woman;
2. Be at least 18 years old;
3. Have experienced SA after the age of 12;
4. Read and speak French;
5. Have adequate Internet access; and f) Present with some post-traumatic stress symptoms (PCL-5 ≥ 10) AND at least mild depressive symptoms (PHQ-9 ≥ 5) AND/OR subclinical insomnia symptoms (ISI ≥ 8).

Exclusion Criteria :

1. Bipolar or psychotic disorder;
2. High suicidal risk, or any other condition requiring immediate intervention;
3. Already benefiting from a psychological intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All persons identifying at least in part with the female gender are included
Enrollment: 204 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder Symptoms | Pre-treatment
  PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - This self-reported questionnaire includes 20 items on a 5-point Likert scale (from 0 = Not at all to 4 = Extremely) evaluating posttraumatic symptoms in the past month. The total score range between 0 and 80 with higher scores indicating higher symptoms severity.
Post-traumatic Stress Disorder Symptoms | Post module (an average of 10 weeks)
  PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - This self-reported questionnaire includes 20 items on a 5-point Likert scale (from 0 = Not at all to 4 = Extremely) evaluating posttraumatic symptoms in the past month. The total score range between 0 and 80 with higher scores indicating higher symptoms severity.
Post-traumatic Stress Disorder Symptoms | 3 months follow-up (12 weeks after last module, which takes on average 30 weeks)
  PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - This self-reported questionnaire includes 20 items on a 5-point Likert scale (from 0 = Not at all to 4 = Extremely) evaluating posttraumatic symptoms in the past month. The total score range between 0 and 80 with higher scores indicating higher symptoms severity.
Depression Symptoms | Pre-treatment
  Patient Health Questionnaire Depression Scale (PHQ-9) - This self-reported questionnaire includes nine items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day). Total severity scores range from 0 to 27, with a higher score indicating a higher severity.
Depression Symptoms | Post module (an average of 10 weeks)
  Patient Health Questionnaire Depression Scale (PHQ-9) - This self-reported questionnaire includes nine items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day). Total severity scores range from 0 to 27, with a higher score indicating a higher severity.
Depression Symptoms | 3 months follow-up (12 weeks after last module, which takes on average 30 weeks)
  Patient Health Questionnaire Depression Scale (PHQ-9) - This self-reported questionnaire includes nine items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day). Total severity scores range from 0 to 27, with a higher score indicating a higher severity.
Insomnia Symptoms | Pre-treatment
  Insomnia Severity Index (ISI) - This self-reported questionnaire includes seven items rated on a 5-point Likert scale (from 0 = No problem to 4 = Very severe problem) that evaluate sleep difficulties in the past two weeks. Total severity scores range from 0 to 28, with a higher score indicating a higher severity of insomnia.
Insomnia Symptoms | Post module (an average of 10 weeks)
  Insomnia Severity Index (ISI) - This self-reported questionnaire includes seven items rated on a 5-point Likert scale (from 0 = No problem to 4 = Very severe problem) that evaluate sleep difficulties in the past two weeks. Total severity scores range from 0 to 28, with a higher score indicating a higher severity of insomnia.
Insomnia Symptoms | 3 months follow-up (12 weeks after last module, which takes on average 30 weeks)
  Insomnia Severity Index (ISI) - This self-reported questionnaire includes seven items rated on a 5-point Likert scale (from 0 = No problem to 4 = Very severe problem) that evaluate sleep difficulties in the past two weeks. Total severity scores range from 0 to 28, with a higher score indicating a higher severity of insomnia.

SECONDARY OUTCOMES:
Sleep quality | Pre-treatment
  Pittsburgh Sleep Quality Index (IQSP)-This self-reported questionnaire evaluating the sleep patterns over the past month. Responses should be the best possible estimates for the majority of days and nights in the last month. Nineteen individual items generate seven component scores, each weighted equally on a 0-3 scale. The sum of the 7 component score yields a total global score, which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality | Post module (an average of 10 weeks)
  Pittsburgh Sleep Quality Index (IQSP)-This self-reported questionnaire evaluating the sleep patterns over the past month. Responses should be the best possible estimates for the majority of days and nights in the last month. Nineteen individual items generate seven component scores, each weighted equally on a 0-3 scale. The sum of the 7 component score yields a total global score, which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality | 3 months follow-up (12 weeks after last module, which takes on average 30 weeks)
  Pittsburgh Sleep Quality Index (IQSP)-This self-reported questionnaire evaluating the sleep patterns over the past month. Responses should be the best possible estimates for the majority of days and nights in the last month. Nineteen individual items generate seven component scores, each weighted equally on a 0-3 scale. The sum of the 7 component score yields a total global score, which has a range of 0-21; higher scores indicate worse sleep quality.
Nightmares | Pre-treatment
  Nightmares Distress Questionnaire (NDQ)- This self-reported questionnaire includes 13 items on a 7-points Likert scale (1= Always to 4= Never) evaluating distress associated with nightmares. A higher score indicates a more severe distress due to nightmares.
Nightmares | Post module (an average of 10 weeks)
  Nightmares Distress Questionnaire (NDQ)- This self-reported questionnaire includes 13 items on a 7-points Likert scale (1= Always to 4= Never) evaluating distress associated with nightmares. A higher score indicates a more severe distress due to nightmares.
Nightmares | 3 month follow-up (12 weeks after last module, which takes on average 30 weeks)
  Nightmares Distress Questionnaire (NDQ)- This self-reported questionnaire includes 13 items on a 7-points Likert scale (1= Always to 4= Never) evaluating distress associated with nightmares. A higher score indicates a more severe distress due to nightmares.
Anxiety Symptoms | Pre treatment
  Generalized Anxiety Disorder Scale (GAD-7) - This self-reported questionnaire includes 7 items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day) evaluating anxiety symptoms in the past two weeks. The total score range between 0 and 21 with higher scores indicating higher symptoms severity.
Anxiety Symptoms | Post module (an average of 10 weeks)
  Generalized Anxiety Disorder Scale (GAD-7) - This self-reported questionnaire includes 7 items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day) evaluating anxiety symptoms in the past two weeks. The total score range between 0 and 21 with higher scores indicating higher symptoms severity.
Anxiety Symptoms | 3 months follow-up (12 weeks after last module, which takes on average 30 weeks)
  Generalized Anxiety Disorder Scale (GAD-7) - This self-reported questionnaire includes 7 items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day) evaluating anxiety symptoms in the past two weeks. The total score range between 0 and 21 with higher scores indicating higher symptoms severity.
Rape Attribution | Pre-treatment
  Rape Attribution Questionnaire (French version)-This questionnaire includes a 25 items on a 5-points Likert scale (1= Never to 5= Very often) evaluating participants' beliefs in the past month about the aggression they experienced.
Rape Attribution | Post- CT module (an average of 5 weeks)
  Rape Attribution Questionnaire (French version)-This questionnaire includes a 25 items on a 5-points Likert scale (1= Never to 5= Very often) evaluating participants' beliefs in the past month about the aggression they experienced.
Maladaptive Beliefs | Pre-treatment
  Posttraumatic Maladaptive Beliefs Scale (French version - under validation)-This self-reported questionnaire includes 14 items on a 7-points Likert scale (1= Completely false to 7= Completely true) evaluating post traumatic maladaptive beliefs of participants.
Maladaptive Beliefs | Post- CT module (an average of 5 weeks)
  Posttraumatic Maladaptive Beliefs Scale (French version - under validation)-This self-reported questionnaire includes 14 items on a 7-points Likert scale (1= Completely false to 7= Completely true) evaluating post traumatic maladaptive beliefs of participants.
Acceptability E-Scale | Post last module (an average of 30 weeks)
  This self-reported questionnaire includes 6 items on a 4-point Likert scale (1= Not at all to 4= a lot) evaluating participant satisfaction with the online intervention.
Appreciation of the online intervention | Post last module (an average of 30 weeks)
  Atrakdiff 2 (RESILIENT platform)-This self-reported questionnaire is a 21 items on a semantic differentiator scale where participants choose words that are closer to their perception of the online intervention among a list of contrasting adjectives.
Semi-structured qualitative interview | Post last module (an average of 30 weeks)
  This semi-structured interview evaluate participants' appreciation of the online platform. The interviewer must ensure that the interview does not exceed 30 minutes and that the content of the interview is limited to the proposed themes. However, the interviewer may modify the questions, add sub-questions and change the order of the questions in order to meet the objectives of the study and to adapt to each participant's speech.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Belleville, Ph.D., Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linde K, Sigterman K, Kriston L, Rucker G, Jamil S, Meissner K, Schneider A. Effectiveness of psychological treatments for depressive disorders in primary care: systematic review and meta-analysis. Ann Fam Med. 2015 Jan-Feb;13(1):56-68. doi: 10.1370/afm.1719. PMID 25583894
- [Background] Bambling, M., et al. (2008).
- [Background] Cook JE, Doyle C. Working alliance in online therapy as compared to face-to-face therapy: preliminary results. Cyberpsychol Behav. 2002 Apr;5(2):95-105. doi: 10.1089/109493102753770480. PMID 12025884
- [Background] Jagger F. The export boning and cutting plant. Vet Rec. 1972 Dec 16;91(25):626-9. doi: 10.1136/vr.91.25.626. No abstract available. PMID 4651423